CLINICAL TRIAL: NCT06653556
Title: An Open-label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LCAR-AIO for the Treatment of Relapsed/Refractory Systemic Lupus Erythematosus (r/r SLE)
Brief Title: A Study of LCAR-AIO in Subjects With Relapsed/Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry); Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Qiubai Li, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2305-0001
Record Dates: First submitted 2024-10-11; First posted 2024-10-22 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Refractory pulmonary Hypertension (PAH); Recurrent/refractory autoimmune hemolytic anemia (r/r AIHA); Recurrent/refractory lupus nephritis (r/r LN)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Hypertension, Pulmonary; Recurrence; Anemia, Hemolytic, Autoimmune; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-AIO T Cells (Experimental): Experimental: Chimeric antigen receptor T cells (LCAR-AIO)
  Each subject will be given a single-dose LCAR-AIO cells infusion at each dose level
  Interventions: Biological: LCAR-AIO T cells

INTERVENTIONS:
Biological: LCAR-AIO T cells — Before treatment with LCAR-AIO T cells, subjects will receive a conditioning regimen.

SUMMARY:
This is a prospective, single-arm, open-label, dose-exploration and expansion clinical study of LCAR-AIO in adult subjects with relapsed/refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label exploratory clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy profiles of LCAR-AIO, a chimeric antigen receptor (CAR) -T cell therapy in subjects with relapsed/refractory systemic lupus erythematosus. Patients who meet the eligibility criteria will receive LCAR-AIO infusion. The study will include the following sequential stages: screening, apheresis, pre-treatment (cell product preparation: lymphodepleting chemotherapy), treatment (LCAR AIO infusion) and follow-up.

ELIGIBILITY:
1. Subjects voluntarily participate in clinical research.
2. Age 18-65 years.
3. Have been diagnosed of SLE at least 6 months before screening.
4. At screening, antinuclear antibody, and/or anti-dsDNA antibody, and/or anti-Sm antibody should be positive.
5. Fulfill relapsed/refractory SLE conditions.
6. Adequate organ function at screening.
7. Clinical laboratory values meet criteria at screening.

Exclusion Criteria:

1. Active infections such as hepatitis and tuberculosis.
2. Other autoimmune diseases.
3. Serious underlying diseases such as tumor, uncontrolled diabetes.
4. Female subjects who were pregnant, breastfeeding, or planning to become pregnant while participating in this study or within 1 year of receiving LCAR-AIO treatment.
5. Participated in other clinical trials within

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Incidence of dose-limiting toxicity (DLT) | 30 days after LCAR-AIO infusion (Day 1)
  DLTs are severe adverse events refers to any untoward medical occurred in a subject participated in a clinical investigation, which have a causal relationship with the treatment and will limit the dose escalation.
Pharmacokinetics in peripheral blood | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  CAR positive T cells levels in peripheral blood after LCAR-AIO infusion.
Recommended Phase 2 Dose (RP2D) regimen finding | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  RP2D established through dose exploratory.

SECONDARY OUTCOMES:
Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  The SELENA-2K scale is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with lupus. A patient's SELENA-2K total score is the sum of all marked lupus related descriptors (seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, hematuria, proteinuria, pyuria, new rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, increased DNA binding, fever, thrombocytopenia, leukopenia). A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Change in Physician global assessment (PGA) scores from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  The physician will place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (Score 0) represents "no activity", and the right-hand boundary (score 3) represents "the most severe activity".
Lupus Low Disease Activity State (LLDAS) response rates at multiple visits post-infusion | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  Percentage of participants achieving the LLDAS. The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. The LLDAS response criteria were: (1) SLEDAI-2K <=4, with no activity in major organ systems (Central nervous system, vascular, renal, cardiorespiratory and constitutional); where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0. (2) no new features of lupus disease activity compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0; (3) Physician global assessment (PGA) (score 0-3), <=1; (4) current prednisolone (or equivalent) dose <=7.5 mg dailyultiple visits.
24h urinary protein/urine protein-to-creatinine ratio (UPCR) changes from baseline up to 104 weeks | Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  Proteinuria will be assessed in lupus nephritis patients basing on 24h urinary protein/UPCR at multiple visits.
Changes from baseline in immunological markers and Immunogenicity (anti-drug antibody) | Time Frame: Minimum 104 Weeks after LCAR-AIO infusion (Day 1)
  Detection of Immunoglobulins, anti-drug antibodies (anti-dsDNA antibody, anti-Sm antibody, etc.) and anti-drug antibody.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No